CLINICAL TRIAL: NCT03347864
Title: Diagnostic Performance of 68Gallium-labeled NOTA-RM26 PET/CT in Breast Tumor Patients
Brief Title: 68Ga-NOTA-RM26 PET/CT in Breast Tumor Patients
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PekingUMCH-NM15
Record Dates: First submitted 2017-11-16; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Breast Tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — 68Ga-NOTA-RM26

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-NOTA-RM26 PET/CT (Experimental): The patients were injected with 1.85 MBq per kilogram body weight of 68Ga-NOTA-RM26 in one dose intravenously and underwent PET/CT scan 30-45 min later
  Interventions: Drug: 68Ga-NOTA-RM26

INTERVENTIONS:
Drug: 68Ga-NOTA-RM26 — 1.85 MBq per kilogram body weight of 68Ga-NOTA-RM26 were injected into the patients before the PET/CT scans

SUMMARY:
This is an open-label positron emission tomography/computed tomography(PET/CT) study to investigate the diagnostic performance and evaluation efficacy of 68Ga-NOTA-RM26 in breast tumor patients. 1.85 MBq per kilogram body weight of 68Ga-NOTA-RM26A will be injected intravenously. Visual and semiquantitative method will be used to assess the PET/CT images.

DETAILED DESCRIPTION:
The gastrin-releasing peptide receptor (GRPR), also known as bombesin receptor subtype II (BB2), is a member of the G protein-coupled receptor family of bombesin receptors. GRPR is over-expressed in various types of human tumors including breast cancer. RM26, a GRPR antagonist with high affinity, was discovered by peptide backbone modification of bombesin analogues.To target gastrin-releasing peptide receptor in neoplastic cells of human breast cancer, peptide NOTA-RM26 was synthesized with a PEG3 linker between NOTA and RM26, and then labeled with 68Ga. An open-label whole-body PET/ CT study was designed to assess its clinical diagnostic value in patients with breast tumor.

ELIGIBILITY:
Inclusion Criteria:

* patients in suspicion of breast cancer by mammography or ultrasonography,and being able to provide basic information and sign the written informed consent form

Exclusion Criteria:

* The exclusion criteria included claustrophobia, pregnancy, breastfeeding, kidney or liver failure, inability to fulfill the study, and undergoing any preceding local or systemic therapies that might interfere with GRPR binding

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value of 68Ga-NOTA-RM26 in breast tumor | 1 year
  The semiquantitative analysis will be performed by the same person for all the cases, and the standardized uptake value (SUV) of the tracer in breast tumor will be measured.

SECONDARY OUTCOMES:
Adverse events collection | 1 week
  Adverse events within 1 week after the injection and scanning of patients and patients will be followed and assessed

CONTACTS AND LOCATIONS:
Overall Officials: Zhaohui Zhu, MD,PHD, Study Chair — Peking Union Medical College Hospital, Chinese Academy of Medical Science and Peking Union Medical College
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China